CLINICAL TRIAL: NCT07248826
Title: Study Protocol for Developing a Methodological Framework and a Theory-informed Dissemination Plan for Herb-drug Interactions-related Clinical Practice Guidelines: a Delphi Survey and a Semi-structured Interview Study
Brief Title: Developing a Methodological Framework and a Dissemination Plan for Herb-drug Interactions-related Clinical Practice Guidelines
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Chinese Medicine Development Fund (Unknown); Chinese Medicine Hospital, Hong Kong Baptist University (Unknown); Hong Kong Poison Control Center, Hospital Authority (Unknown); Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Principal Investigator, Yin Ting Cheung, Associate Professor, Chinese University of Hong Kong
Other Study IDs: SBRE-25-0100
Record Dates: First submitted 2025-11-17; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-08

CONDITIONS: Herb-drug Interactions
Keywords: herb-drug interactions; methodological framework; evidence-based approach; Delphi method; dissemination plan; semi-structured interview

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Delphi Panel: The expert panel with the following backgrounds will be invited to participate in the Delphi survey: a. registered Chinese medicine practitioners, herbalists, or researchers in the field of integrated Chinese and Western medicine; b. physicians providing care in integrated Chinese and Western medicine settings; c. healthcare administrators or policymakers from clinics/hospitals directly involved in developing or reviewing clinical practice guidelines related to integrated Chinese and Western medicine.
  Interventions: Other: Delphi method survey
- Participants of semi-structured interview: Experts with the following backgrounds will be invited to participate in the semi-structured interview: a. registered Chinese medicine practitioners, herbalists, or researchers in the field of integrated Chinese and Western medicine; b. physicians providing care in integrated Chinese and Western medicine settings; c. healthcare administrators or policymakers from clinics/hospitals directly involved in developing or reviewing clinical practice guidelines related to integrated Chinese and Western medicine.
  Interventions: Other: Semi-structured interview

INTERVENTIONS:
Other: Delphi method survey — The Delphi survey intervention will comprise two rounds of structured questionnaire surveys to gather stakeholder consensus on the factors and components to consider when translating herb-drug interactions' evidence into recommendations. Following the first round of surveys, we will calculate the median score and interquartile range for each consideration factor, expressing participant consensus on these factors as percentages. Consideration factors achieving consensus in the first round will be considered for inclusion in the clinical practice guideline development framework. For factors where consensus was not reached, we will summarize relevant opinions and further evaluate them in the second round of the Delphi survey. Finally, descriptive statistics (frequencies and proportions) will be used to summarize the quantitative results of the Delphi survey.
  Groups: Delphi Panel
Other: Semi-structured interview — A face-to-face semi-structured interview with participants will be conducted. Interview questions will be developed based on the Theoretical Domains Framework (TDF). The interview will cover three main aspects: a. participants' experiences in searching for evidence and clinical practice guidelines (CPGs) related to herb-drug interactions (HDIs); b. barriers and facilitators encountered when retrieving HDI-related CPGs or obtaining information from existing CPGs; c. their views on the ideal platform for disseminating HDI-related CPGs.
  Groups: Participants of semi-structured interview

SUMMARY:
The goal of this observational study is to develop a methodological framework for clinical practice guidelines (CPGs) related to herb-drug interactions (HDIs). It will also learn barriers and facilitators of disseminating HDI-related CPGs and formulate a dissemination plan. The main questions it aims to answer are:

1. develop a methodological framework for HDI-related CPGs using a Delphi method;
2. identity barriers and facilitators of disseminating HDI-related CPGs through semi-structured interviews and formulate a theory-informed dissemination plan to promote the uptake of CPGs locally and internationally.

   * Participants in the Delphi survey will engage in a consensus development to determine the framework of HDI-related CPGs, including key characteristics and components of this framework.
   * Participants in the semi-structured interviews will be interviewed on the following topics: their experiences in searching for evidence and CPGs related to HDIs; barriers and facilitators encountered when obtaining information from existing CPGs; their views on the ideal platform for disseminating HDI-related CPGs.

DETAILED DESCRIPTION:
In recent decades, the combined use of conventional (Western) drugs and herbal medicines has become increasingly common. Numerous studies have reported the prevalence of combined use, ranging from approximately 14% to 45%. The prevalence may be higher in low- and middle-income countries (LIC/LMIC), as studies have indicated that Traditional and Complementary Medicine is more popular in these regions, with Palestine and China reporting the highest prevalence of herbal medicine use. Although the initial purpose of combining conventional drugs and herbal medicines is to improve health and reduce adverse reactions, these combinations may yield either beneficial or harmful interactions. Herb-drug interactions (HDIs) can occur at pharmacokinetic (PK) and pharmacodynamic (PD) levels. PK interactions are those that affect the processes of drug absorption, distribution, metabolism, or excretion (known as ADME interactions). For example, St. John's Wort can reduce plasma concentrations of concomitantly administered CYP3A substrates such as alprazolam by inducing CYP3A4 activity. PD interactions are those in which the effect of one drug is altered by the presence of another drug at its site of action. For instance, ginkgo combined with anticoagulants such as warfarin can produce an additive effect, increasing the risk of bleeding. A scoping review focusing on cancer patients estimated that approximately 45.4% of patients using herbal medicines were at risk of harmful HDIs, which can cause adverse reactions and even pose a threat to people's lives. Therefore, it is essential to prioritize safety alongside efficacy of integrated therapies.

I. Gaps in HDI-related clinical practice guidelines (CPGs) The World Health Organization (WHO), U.S. Food and Drug Administration (FDA), and European Medicines Agency (EMA) have issued technical documents and established regulatory frameworks to support safe concurrent use of conventional drugs and herbal medicines. However, these efforts have not led to a proliferation of HDI-related CPGs. HDI-related CPGs remain scarce. Existing CPGs normally lack specific management and monitoring strategies and may not be well aligned with real-world practice, limiting their utility for clinicians. For example, a 2001 guideline recommended avoiding the combined use of Korean Ginseng and Warfarin unless under medical supervision, without specifying the type of supervision required. Furthermore, information provided by existing clinical decision support systems is inconsistent, creating further challenges on implementation in this area. A study reported significant discrepancies in the direction and severity of interactions between warfarin and medicinal plants across four commonly used online clinical decision resources, which could compromise clinical decision-making.

Beyond these gaps, there is currently no methodological framework existing for translating HDI evidence into implementable CPGs. Although there are frameworks such as GRADE Evidence to Decision (EtD) assisting in synthesizing evidence into recommendations, they are primarily designed for interventions with clearly defined PICO questions. This intervention-oriented nature limits their applicability to HDI, where herbal medicines represent complex, heterogeneous exposures rather than standardized interventions. Therefore, it is urgent to develop a dedicated framework for HDI-related CPGs to bridge evidence and practice.

II. Gaps in dissemination of HDI-related CPGs Integrating CPG recommendations into clinical practice is often slow and challenging, with an average lag of 17 years for evidence to influence routine care. To mitigate time lag, dissemination planning should begin alongside CPG development, as recommended by the Scottish Interprofessional Guidelines Network (SIGN). Several guideline dissemination platforms, including MAGIC, ECRI Guidelines Trust, and the Guidelines International Network, have been developed to organize fragmented evidence or recommendations into structured, searchable, and updatable formats to facilitate adoption. However, these platforms are limited by narrow scope and poor accessibility, and often rely on external links. In the context of HDIs, clinicians often access information through software and online resources, yet encounter conflicting data, insufficient detail, and usability challenges. Patients also express a desire for reliable HDI information. Despite this demand, few studies have investigated barriers, facilitators or end-user preferences for disseminating HDI-related CPGs. Addressing these gaps is essential to improve the accessibility, clarity and uptake of HDI-related CPGs.

To address the scarcity of HDI-related CPGs and the lack of effective dissemination strategies, the specific objectives of this study are to:

i. develop a methodological framework for HDI-related CPGs through a modified Delphi method informed by findings from a scoping review; and ii. identity barriers to and facilitators of disseminating HDI-related CPGs, as well as end-user preferences through semi-structured interviews, and then design a theory-informed dissemination plan to promote uptake of CPGs internationally.

ELIGIBILITY:
Inclusion Criteria:

* Registered Chinese medicine practitioners, herbalists, or researchers in the field of integrated Chinese and Western medicine;
* or physicians providing care in integrated Chinese and Western medicine settings;
* or healthcare administrators or policymakers from clinics/hospitals directly involved in developing or reviewing clinical practice guidelines related to integrated Chinese and Western medicine.

Exclusion Criteria:

* Panelists who are unable to commit to participating in all rounds of the Delphi process;
* or panelists who are unable to complete the online questionnaire in either Chinese or English;
* or panelists who are unable to conduct the interview in either English or Cantonese.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population encompass a diverse group of experts, including registered Chinese medicine practitioners, herbalists, or researchers; clinicians; and healthcare administrators or policymakers in the field of integrated Chinese and Western medicine. This expert panel aims to gather a broad range of perspectives to ensure the establishment of a comprehensive and standardized framework for developing guidelines on herb-drug interactions.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Degree of consensus | Through study completion, an average of 6 months
  The level of agreement for all statements achieving consensus among the expert panel. This study sets the consistency threshold at 75%. Namely, if more than 75% of participants select either "Relevant" or "Highly relevant", the item will be considered to have reached consensus for inclusion in the final framework. Conversely, if more than 75% of participants select either "Highly irrelevant" or "Irrelevant", the item will be considered to have reached consensus for exclusion. Items that do not meet either criterion will be considered as failing to reach consensus and be carried forward to the next round.
Experiences in searching for clinical practice guidelines (CPGs) related to herb-drug interactions (HDIs); barriers and facilitators encountered during retrieving process; views on the ideal platform for disseminating HDI-related CPGs and the framework | Through study completion, an average of 6 months
  The primary outcome will be assessed by asking participants about the sources they refer to for recommendations on HDIs; what barriers or facilitators they encountered when retrieving HDI-related CPGs; what factors will promote or hinder the development of HDI-related CPGs or the CPG dissemination platform; what anticipated benefits or potential traps the development of the CPG dissemination platform might bring; and the target audience, ideal dissemination channels, etc.

REFERENCES:
- [Background] Lam CS, Koon HK, Ma CT, Au KY, Zuo Z, Chung VC, Cheung YT. Real-world data on herb-drug interactions in oncology: A scoping review of pharmacoepidemiological studies. Phytomedicine. 2022 Aug;103:154247. doi: 10.1016/j.phymed.2022.154247. Epub 2022 Jun 7. PMID 35716539
- [Background] Fugh-Berman A. Herb-drug interactions. Lancet. 2000 Jan 8;355(9198):134-8. doi: 10.1016/S0140-6736(99)06457-0. PMID 10675182
- [Background] Wong CHL, Wu IXY, Adams J, Steel A, Wardle J, Wu JCY, Leung TH, Chung VCH. Development of Evidence-Based Chinese Medicine Clinical Service Recommendations for Cancer Palliative Care Using Delphi Approach Based on the Evidence to Decision Framework. Integr Cancer Ther. 2020 Jan-Dec;19:1534735420940418. doi: 10.1177/1534735420940418. PMID 32646246
- [Background] Zuo Z, Huang M, Kanfer I, Chow MS, Cho WC. Herb-drug interactions: systematic review, mechanisms, and therapies. Evid Based Complement Alternat Med. 2015;2015:239150. doi: 10.1155/2015/239150. Epub 2015 Feb 22. No abstract available. PMID 25792995
- [Background] Bush TM, Rayburn KS, Holloway SW, Sanchez-Yamamoto DS, Allen BL, Lam T, So BK, Tran de H, Greyber ER, Kantor S, Roth LW. Adverse interactions between herbal and dietary substances and prescription medications: a clinical survey. Altern Ther Health Med. 2007 Mar-Apr;13(2):30-5. PMID 17405676